CLINICAL TRIAL: NCT02403102
Title: Imageguided Theranostics in Multiple Myeloma
Acronym: iTIMM
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); National Institute for Health Research, United Kingdom (Other Government); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: 15/LO/0036 CCR4236
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2022-12-14 (Actual); Status verified 2021-05

CONDITIONS: Cancer; Myeloma
Keywords: Magnetic Resonance Imaging; Myeloma; Autograft
MeSH Terms: conditions — Neoplasms; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients who undergo autograft have regular blood tests and marrow sampling and we will use these samples, to look at other factors which influence patient outcomes such as genetics, without compromising routine care. Some of the genetic tests performed on the bone marrow are not routine so we will obtain additional consent to do this.
Oversight: Data Monitoring Committee: No

SUMMARY:
Theranostics is the use of a diagnostic test to decide which patients will benefit from a certain treatment.

The current standard treatment for patients with myeloma is induction chemotherapy followed by peripheral stem cell transplant. Although there are options for timing of treatments, patient outcomes are variable and the investigators do not currently know which patients benefit from which treatment schedule. There is evidence to suggest that residual disease on imaging after treatment is an indicator for a worse prognosis, however the best time point for this imaging is currently not known. This study is designed to show if there is an optimum time point for correlation between imaging and prognosis.

Several studies have indicated that MRI is better at detecting disease than FDG PET/CT and the investigators will confirm this when patients are first diagnosed, by performing both FDG PET/CT and whole body diffusion weighted MRI.

Patients will then be followed up with whole body diffusion weighted MRI after induction chemotherapy and 3 months post autograft. The investigators will look at the amount of disease present on these scans and correlate this with outcomes.

There are likely to be other factors which influence patient outcomes (such as genetics) and the investigators will also look at some of these. Patients who undergo autograft have regular blood tests and marrow samples taken as part of routine care, the investigators will use some of these samples (without compromising the patients treatment) to analyses some of these other factors. If the investigators are able to determine a correlation of genetic factors with outcome this information could be used in future research.

Theranostics is the use of a diagnostic test to decide which patients will benefit from a certain treatment.

The current standard treatment for patients with myeloma is induction chemotherapy followed by peripheral stem cell transplant. Although there are options for timing of treatments, patient outcomes are variable and the investigators do not currently know which patients benefit from which treatment schedule. There is evidence to suggest that residual disease on imaging after treatment is an indicator for a worse prognosis, however the best time point for this imaging is currently not known. This study is designed to show if there is an optimum time point for correlation between imaging and prognosis.

Several studies have indicated that MRI is better at detecting disease than FDG PET/CT and the investigators will confirm this when patients are first diagnosed, by performing both FDG PET/CT and whole body diffusion weighted MRI.

Patients will then be followed up with whole body diffusion weighted MRI after induction chemotherapy and 3 months post autograft. The investigators will look at the amount of disease present on these scans and correlate this with outcomes.

There are likely to be other factors which influence patient outcomes (such as genetics) and the investigators will also look at some of these. Patients who undergo autograft have regular blood tests and marrow samples taken as part of routine care, the investigators will use some of these samples (without compromising the patients treatment) to analyses some of these other factors. If the investigators are able to determine a correlation of genetic factors with outcome this information could be used in future research.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 with multiple myeloma planned for autograft.

Exclusion Criteria:

* MRI incompatible metal implants
* Claustrophobia
* Diagnosis of other malignancy within 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myeloma planned for autograft.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Construct a ROC curve and calculate area under the curve (AUC) to show that the burden of disease at 3 months post autograft (WB-DWI score) is predictive of disease status at 2 years. | 2 years post autograph

SECONDARY OUTCOMES:
Use multivariate/univariate analysis to identify the best single or combination MRI parameter(s) to predict disease status at 2 years | 2 years post autograph
Identify optimal cut-off point with best sensitivity and specificity to predict disease status at 2 years. | 2 years post autograph
Calculate PFS for patients grouped by optimal cut-off. | 2 years post autograph
Overall survival (OS) in patients with residual disease on WB-DWI post induction and 3 months post autograft. | 2 years post autograph

CONTACTS AND LOCATIONS:
Overall Officials: Christina Messiou, Dr, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Messiou C, Porta N, Sharma B, Levine D, Koh DM, Boyd K, Pawlyn C, Riddell A, Downey K, Croft J, Morgan V, Stern S, Cheung B, Kyriakou C, Kaczmarek P, Winfield J, Blackledge M, Oyen WJG, Kaiser MF. Prospective Evaluation of Whole-Body MRI versus FDG PET/CT for Lesion Detection in Participants with Myeloma. Radiol Imaging Cancer. 2021 Sep;3(5):e210048. doi: 10.1148/rycan.2021210048. PMID 34559006